CLINICAL TRIAL: NCT02267876
Title: Longitudinal Clinical Evaluation of the HPV Assay on the BD VIPER LT System With Cervical Specimens
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: BDS-USLHPV
Record Dates: First submitted 2014-10-14; First posted 2014-10-20 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Cervical Neoplasms; Human Papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BD VIPER LT
  Interventions: Device: BD HPV Assay on Viper LT; Procedure: Colposcopy

INTERVENTIONS:
Device: BD HPV Assay on Viper LT — The BD HPV specimen will be tested with the BD HPV Assay on the Viper LT instrument.
Procedure: Colposcopy — The colposcopy will be performed on subjects that have abnormal cytology. At the third year visit all subjects will have an exit colposcopy.

SUMMARY:
The purpose of the study is to assess the cumulative disease detection of greater than or equal to Cervical intraepithelial neoplasia 2 (CIN2) and greater than or equal to Cervical intraepithelial neoplasia 3 (CIN3) in the subjects over 3 years using the subject's HPV status and cytology status from the BDS-USHPV baseline results

ELIGIBILITY:
Inclusion Criteria:

* Subject enrolled into the protocol BDS-USHPV and identified as eligible for the longitudinal protocol • Subjects enrolled into protocol BDS-USHPV with a baseline colposcopy and biopsy procedure and not treated.

Exclusion Criteria:

* Subjects with prior complete or partial hysterectomy involving removal of the cervix
* Subjects on whom conization, LEEP, cervical laser surgery, or cryosurgery has been performed since enrollment into the BDS-USHPV study
* Year 3 visit can not exceed 3 years and 6 months from the baseline visit

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were selected from a baseline study BDS-USHPV, which included female healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 6730 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Cumulative risk of Cervical Intraepithelial Neoplasia 2 and 3 (CIN2 and CIN3) over three years in Human Papillomavirus (HPV) Positive Patients. | 3 years
  Cumulative risk is a measure of the total risk that a certain event will happen during a given period of time. In this longitudinal study, it refers to the risk of developing >=CIN2 or >=CIN3 in subjects over a three year period using the subjects' HPV status at baseline versus cytology status at baseline.
Absolute Risk of Cervical Intraepithelial Neoplasia 2 and 3 (CIN2 and CIN3) over 3 years in Human Papillovirus (HPV) Positive Patients. | 3 years
  Absolute risk will be calculated as: (number of disease cases)/(number of patients at risk).
To evaluate different screening strategies using Human Papillovirus (HPV) results with 16/18/45 genotyping and cytology. | 3 years
  The sensitivity and specificity of HPV primary screening algorithms for identifying ≥ CIN2 and ≥ CIN3 using genotyping and cytology will be calculated.

SECONDARY OUTCOMES:
Cumulative Risk of Cervical Intraepithelial Neoplasia 2 and 3 (CIN2 and CIN3) over 3 years in NILM (Negative for Intraepithelial lesion or malignancy) cytology and Human Papillovirus (HPV) Negative Patients. | 3 years
  Cumulative risk is a measure of the total risk that a certain event will happen during a given period of time. In this longitudinal study, it refers to the risk of developing >=CIN2 or >=CIN3 over a three year period for the population of women negative for intraepithelial lesions or malignancy (NILM) cytology and with Human Papillovirus (HPV) negative results.
Absolute Risk of Cervical Intraepithelial Neoplasia 2 and 3 (CIN2 and CIN3) over 3 years in NILM (Negative for Intraepithelial Lesion or Malignancy) cytology and Human Papillomavirus (HPV) Negative Patients. | 3 years
  Absolute risk will be calculated as: (number of disease cases)/(number of patients at risk).
Evaluate Different Screening Strategies Using HPV Results with Genotyping (other than 16/18/45) and Cytology. | 3 years
  The sensitivity and specificity of HPV primary screening algorithms for identifying ≥ CIN2 and ≥ CIN3 using genotyping and cytology will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Tobi Karchmer, MD, Study Director — Becton, Dickinson and Company
Locations (40):
- United States (39):
  - University of Alabama, Birmingham, Alabama
  - Mobile OB/GYN, Mobile, Alabama
  - Women's Health Research of Arizona, Phoenix, Arizona
  - Quality of Life Medical & Research Center, Tucson, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Women's Health Care Research Corp., San Diego, California
  - Blueskies Center for Women, Colorado Springs, Colorado
  - Health Awareness Inc., Jupiter, Florida
  - Altus Research, Lake Worth, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Comprehensive Clinical Trails, LLC, West Palm Beach, Florida
  - Medical Network for Education & Research, Decatur, Georgia
  - Fellows Research Alliance - Savannah, Savannah, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Indiana University, Indianapolis, Indiana
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Louisiana State University, New Orleans, Louisiana
  - BD 54 Loveton, Sparks, Maryland
  - Saginaw Valley Medical Research, Saginaw, Michigan
  - Virtua Phoenix OB/GYN, Moorestown, New Jersey
  - Meridian Health / Jersey Shore University Medical Center, Neptune City, New Jersey
  - Quest Laboratories, Teterboro, New Jersey
  - TriCore, Albuquerque, New Mexico
  - Research Pathology Associates, LLC, Irvington, New York
  - Montefiore Medical Center, The Bronx, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - HWC Women's Research Center, Englewood, Ohio
  - Center for Women's Health of Lansdale, Lansdale, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Reading Health Physician Network, West Reading, Pennsylvania
  - Fellows Research Alliance - Bluffton, Bluffton, South Carolina
  - James T. Martin Jr. OB/GYN, North Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Center for Disease Detection, LLC, San Antonio, Texas
  - Physicians Research Options, Draper, Utah
  - Research Pathology Associates, Charlottesville, Virginia
  - Tidewater Clinical Research, Virginia Beach, Virginia
- BioVision, Montreal, Quebec, Canada